CLINICAL TRIAL: NCT00701064
Title: Bright Light: An Adjunct Treatment for Combat PTSD
Brief Title: Bright Light: An Adjunct Treatment for Combat Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-008-08S
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; phototherapy; anxiety; depression; sleep; negative ion generator
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bright Light Exposure (Experimental): Bright Light (30 min/day)
  Interventions: Other: Bright Light Exposure
- Negative Ion Generator (Placebo Comparator): Negative Ion Generator (30 min/day)
  Interventions: Other: Negative Ion Generator

INTERVENTIONS:
Other: Bright Light Exposure — Administered via bright light box
  Arms: Bright Light Exposure
Other: Negative Ion Generator — Administered via Negative Ion Generatore
  Arms: Negative Ion Generator

SUMMARY:
The investigators are testing novel treatments for combat PTSD: bright light exposure and negation ion exposure.

DETAILED DESCRIPTION:
Seventy Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans with posttraumatic stress disorders (PTSD) will be randomly assigned to one of two 4-week treatments (45 min/day): (1) bright light exposure or (2) a negative ion generator. Clinical assessments ,as well as self-reported measures of PTSD, anxiety, depression, and sleep will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Veteran of Operation Iraqi Freedom or Operation Enduring Freedom with Posttraumatic Stress Disorder
* receiving other treatment or stopped other treatment prior to study

Exclusion Criteria:

* bipolar disorder
* psychosis
* alcohol/drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2012-11-21 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D. Youngstedt, PhD, Principal Investigator — Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC
Locations (1):
- Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bright Light Exposure | Negative Ion Generator
Started | 35 | 36
Completed | 31 | 32
Not Completed | 4 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — initiated other PTSD treatment | 2 | 2

BASELINE CHARACTERISTICS:
Population: Veterans with PTSD
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright Light Exposure | Negative Ion Generator | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (9.3) | 36.0 (8.0) | 36.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 27 | 28 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 21 | 23 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 36 | 71
Clinician Administered PTSD Scale (CAPS2) [Mean (Standard Deviation); unit: units on a scale] — PTSD assessed by a skilled clinician, the CAPS2 is the most common clinical and experimental measure of PTSD severity. It is designed to assess changes in PTSD severity over time, the scale ranges from 0-136. Higher levels indicate greater severity of PTSD. Scores of 30 or more or 40 or more have been considered indicated of moderate severity PTSD.
  units on a scale | 63.0 (20.2) | 62.3 (26.6) | 62.6 (23.5)
Clinical Global Impression Scale (CGI) [Mean (Standard Deviation); unit: units on a scale] — Clinical judgement of the severity of one's condition at baseline (7 point scale: 1=normal; 4=moderately ill; 7= among the most severely ill)
  units on a scale | 4.3 (0.9) | 4.2 (1.6) | 4.3 (1.3)
PTSD Checklist (PCL) [Mean (Standard Deviation); unit: units on a scale] — A 17-item self-rated PTSD scale ranging from 17-105, with higher levels indicating more severe PTSD. The PCL correlates highly with the CAPS-2.
  units on a scale | 45.3 (10.1) | 47.2 (15.2) | 46.3 (12.9)
Pittsburgh Sleep Quality Inventory [Mean (Standard Deviation); unit: units on a scale] — A common instrument that assesses sleep quality over the previous month. The PSQI range is 0-21 with higher scores indicating worse sleep. Scores of > 5 have been considered indicative of a sleep problem.
  units on a scale | 10.3 (3.4) | 10.4 (4.2) | 10.4 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Assessed PTSD Scale (CAPS-2)
Description: The CAPS-2 is administered by a trained clinician. It is designed to assess changes in PTSD severity over time, the scale ranges from 0-136. Higher levels indicate greater severity of PTSD.
Time Frame: Mean change from baseline to post-treatment (5-6 weeks later)
Population: Separate analysis will be conducted to include drop-outs and exclusions. reported are end of study data
Measure: Mean (Standard Deviation); unit: change in units on scale
Groups:
- Arm 1: Bright Light: Bright Light (30 min/day)
  Bright Light Exposure: Administered via bright light box
- Arm 2: Placebo Negative Ion Generator: Negative Ion Generator (30 min/day)
  Inactivated Negative Ion Generator: Administered via Negative Ion Generator
Arm/Group | Arm 1: Bright Light | Arm 2: Placebo Negative Ion Generator
Number analyzed (Participants) | 31 | 31
change in units on scale | 20.10 (18.63) | 8.84 (17.89)

2. Primary Outcome: Clinical Global Impressions Scale (CGI)
Description: The CGI assesses baseline severity on a 7-point scale, and change on 7-point scale. (1=normal; 4=moderately ill; 7= among the most severely ill). Change: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse
Time Frame: Baseline severity to post-treatment (4 weeks later) Change
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Arm 1: Bright Light | Arm 2: Placebo Negative Ion Generator
Number analyzed (Participants) | 31 | 31
units on scale | 2.61 (0.18) | 3.16 (0.17)

3. Secondary Outcome: Posttraumatic Stress Disorder Checklist (PCL-M)
Description: Self-rated PTSD scale with 17 items (rated 1-5) with range of 17-85. Higher score = worse severity of PTSD. Reported are decreases from baseline to end-of-study.
Time Frame: Baseline to following 4-week treatment
Measure: Mean (Standard Error); unit: decrease in units on scale
Arm/Group | Arm 1: Bright Light | Arm 2: Placebo Negative Ion Generator
Number analyzed (Participants) | 31 | 31
decrease in units on scale | 11.03 (1.93) | 6.25 (1.61)

ADVERSE EVENTS:
Time Frame: At the end of baseline period and weekly during the 4-week intervention, we monitored the subjects for suicidal thoughts with the Beck Suicide Scale.
Groups:
- Arm 1: Bright Light Exposure: Bright Light (30 min/day)
  Bright Light Exposure: Administered via bright light box
- Arm 2: Negative Ion Generator: Negative Ion Generator (30 min/day)
  Negative Ion Generator: Administered via Negative Ion Generatore
Arm/Group | Arm 1: Bright Light Exposure | Arm 2: Negative Ion Generator
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes